CLINICAL TRIAL: NCT04140786
Title: Optimization of Intravenous Gentamicin Treatment to Restore Functional Laminin 332 in JEB Patients With Nonsense Mutations
Brief Title: Optimizing IV Gentamicin in JEB
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, David Woodley, Professor of Dermatology, Keck School of Medicine, University of Southern California
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-19-00760
Record Dates: First submitted 2019-10-23; First posted 2019-10-28 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Junctional Epidermolysis Bullosa
Keywords: Nonsense mutation
MeSH Terms: conditions — Epidermolysis Bullosa, Junctional | interventions — Gentamicins; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daily IV Gentamicin (Experimental): Once daily (for 24 days) IV infusions of 10 mg/kg gentamicin delivered over a 30-60 minute period.
  Interventions: Drug: Gentamicin Sulfate, Injectable
- Biweekly IV Gentamicin (Experimental): Twice weekly (for 3 months or 24 total) IV infusions of 10 mg/kg gentamicin delivered over a 30-60 minute period.
  Interventions: Drug: Gentamicin Sulfate, Injectable

INTERVENTIONS:
Drug: Gentamicin Sulfate, Injectable — 10mg/kg prepared from commercially available stock (typically Kabi Pharmaceuticals) by licensed pharmacists.
  Other Names: Gentamicin, Garamycin

SUMMARY:
Herlitz junctional epidermolysis bullosa (H-JEB), an incurable and fatal inherited skin disease, is caused by loss-of-function mutations in LAMA3, LAMB3 and LAMC2. These mutations result in diminished laminin 332 and epidermal-dermal adherence. 85% of JEB patients have nonsense mutations in LAMA3, LAMB3, or LAMC2, suggesting that H-JEB is a prime therapeutic target for nonsense suppression therapy. The investigators recently demonstrated in three patients that topical gentamicin created new and stable laminin 332 at the dermal-epidermal junction (DEJ), and also improved wound closure and skin quality. Furthermore, these preliminary studies showed that intravenous gentamicin also induced laminin 332 and transiently improved patients' clinical outcomes. No untoward side effects occurred. The investigators propose to optimize the intravenous gentamicin regimen including dosage and infusion schedules to enhance the therapeutic outcome. The milestones will be an increase of laminin 332 in the patients' DEJ, improvement in EB Disease Activity Scores, and no gentamicin-associated side effects.

DETAILED DESCRIPTION:
RATIONALE:

Herlitz junctional epidermolysis bullosa (H-JEB), an incurable and fatal inherited skin disease, is caused by loss-of-function mutations in LAMA3, LAMB3 and LAMC2. These mutations result in diminished laminin 332 and epidermal-dermal adherence. 85% of JEB patients have nonsense mutations in LAMA3, LAMB3, or LAMC2, suggesting that H-JEB is a prime therapeutic target for nonsense suppression therapy. The investigators recently demonstrated in three patients that topical gentamicin created new and stable laminin 332 at the dermal-epidermal junction (DEJ), and also improved wound closure and skin quality. Furthermore, these preliminary studies showed that intravenous gentamicin also induced laminin 332 and transiently improved patients' clinical outcomes. No untoward side effects occurred. The investigators propose to optimize the intravenous gentamicin regimen including dosage and infusion schedules to enhance the therapeutic outcome.

INTERVENTION:

There will be two study designs on JEB patients with nonsense mutation(s):

A. Short Term Daily IV Gentamicin Study: Three patients of any age with JEB caused by nonsense mutation(s) in the LAMA3 and LAMB3 genes will receive intravenous gentamicin (10 mgs/kg) daily for 24 days and then stop. Prior to treatment and at 1 month and 3 months post treatment, selected skin test sites will have skin biopsies and the specimens evaluated for the expression of laminin 332 at the dermal-epidermal junction by direct immunofluorescent staining of the skin. Safety parameters such as physical exam, review of systems, laboratory tests, audiometry, and renal function at the same time periods.

B. Long Term Biweekly IV Gentamicin Study: Three patients of any age with JEB caused by nonsense mutation(s) in the LAMA3 and LAMB3 genes will receive intravenous gentamicin (10 mgs/kg) twice weekly for 3 months (24 total infusions) and then stop. Before and after evaluations will be performed and will be the same as those in the short term intravenous study outlined above.

STUDY POPULATION:

3 adults/children for who have JEB due to nonsense mutations in the LAMA3 or LAMB3 gene for each intervention arm.

STUDY ENDPOINTS OR OUTCOMES Analysis of safety parameters, wound healing, and generation of new laminin 332 at the dermal-epidermal junction of the skin by direct immunofluorescent stain.

FOLLOW-UP Participants will be followed out to 90 days post treatment

STATISTICS Without treatment, these JEB patients have little or no laminin A3/laminin B3/laminin 332 at their dermal-epidermal junction. The expression of any newly generated laminin 332 will be measure against normal human skin (100%) by NIH Image J software.

PLANS FOR ANALYSIS Safety parameters are outlined above and will be examined at baseline and after each patient visit. Efficacy parameters outlined above will be measured at baseline and at post treatment days 30 and 90.

ELIGIBILITY:
Inclusion Criteria:

* JEB patients with nonsense mutations in LAMB3 or LAMA3 in either one or two alleles
* Immunofluorescence (IF) analysis showing absence or decreased laminin 332 expression at their DEJ compared with normal skin.

Exclusion Criteria:

* Pre-existing known auditory impairment.
* Pre-existing known renal impairment.
* Pre-existing known allergies to aminoglycosides or sulfate compounds.
* Pregnancy.
* Recent exposure to systemic gentamicin within the past 6 weeks.
* Current use of any medications with known potential ototoxicity or nephrotoxicity.

Min Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Laminin 332 Expression in Skin | 3 months
  Expression of laminin 332 as assessed by immunofluorescence of patient skin sections as a percentage of normal skin.
Safety (Ototoxicity) | 3 months
  Testing for any gentamicin-associated auditory impairment as assessed by pure-tone audiometry assessments.
Safety (Nephrotoxicity) | 3 months
  Testing for any gentamicin-associated renal impairment as assessed by calculated creatinine clearance.
Safety (Autoimmune Response) | 3 months
  Testing for the presence of auto antibodies to newly formed laminin 332 in response to gentamicin as assessed by specific ELISA.

SECONDARY OUTCOMES:
Wound Healing | 3 months
  Size of skin wounds selected for monitoring at baseline as assessed by computer assisted planimetry of photographs.
Epidermolysis Bullosa Disease and Activity and Scarring Index (EBDASI) | 3 months
  A disease scoring system designed for patients with epidermolysis bullosa (EB).

CONTACTS AND LOCATIONS:
Overall Officials: Mei Chen, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mosallaei D, Hao M, Antaya RJ, Levian B, Kwong A, Cogan J, Hamilton C, Schwieger-Briel A, Tan C, Tang X, Woodley DT, Chen M. Molecular and Clinical Outcomes After Intravenous Gentamicin Treatment for Patients With Junctional Epidermolysis Bullosa Caused by Nonsense Variants. JAMA Dermatol. 2022 Apr 1;158(4):366-374. doi: 10.1001/jamadermatol.2021.5992. PMID 35234826